CLINICAL TRIAL: NCT00689689
Title: A Randomized Clinical Study Comparing a Fully-Coated Cementless Stem Versus a Cemented Stem for Total Hip Replacements
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDHA-RL-005
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2008-05

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fully Coated Prodigy Stem (AML) (Active Comparator): Total hip arthroplasty with fully coated prodigy stem (AML)
  Interventions: Device: Fully coated Prodigy stem
- Cemented Endurance Hip Stem (Active Comparator): Total hip arthroplasty with cemented Endurance hip stem component
  Interventions: Device: Cemented Endurance Stem

INTERVENTIONS:
Device: Fully coated Prodigy stem — Total hip arthroplasty with fully coated Prodigy stem
  Arms: Fully Coated Prodigy Stem (AML)
Device: Cemented Endurance Stem — total hip arthroplasty with cemented endurance stem
  Arms: Cemented Endurance Hip Stem

SUMMARY:
The purpose of this study is to answer the question as to whether or not a fully coated cementless stem is equal to or better than a cemented stem in patients over 72 years with good bone quality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing surgery for total hip replacements, including diagnosis of osteoarthritis, rheumatoid arthritis, traumatic and post-traumatic arthritis, avascular necrosis and congenital dislocation of the hip. Congenital dislocation of the hip will be included where small but anatomical acetabuli are present, ie., the acetabuli located near the tear-drop
* Revisions of failed osteotomies may be included
* Bone quality felt to be acceptable to the surgeon for cementless arthroplasty preoperatively in patients > 72 years of age

Exclusion Criteria:

* Patients with active infection
* Revision cemented total hip replacement
* Charcot joints
* Patients with primary or secondary bone tumors in the vicinity of the joint to be replaced
* C.D.H. with abnormally placed acetabuli or femoral canals
* Fibromyalgia patients

Min Age: 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 1998-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Revision

SECONDARY OUTCOMES:
Womac
SF-12

CONTACTS AND LOCATIONS:
Overall Officials: Ross K Leighton, MD, FRCS(C), Principal Investigator — Capital Health, Canada
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada